CLINICAL TRIAL: NCT01602575
Title: Neuroimaging Biomarkers of Mind-Body Treatment Response in Chronic Visceral Pain
Brief Title: Neuroimaging and Biomarkers in Chronic Visceral Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Kirsten Tillisch, MD, Principal Investigator, University of California, Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R01AT007137 (NIH); R01AT007137 (NIH)
Record Dates: First submitted 2012-05-17; First posted 2012-05-21 (Estimated); Last update posted 2018-05-14 (Actual); Status verified 2018-05

CONDITIONS: Irritable Bowel Syndrome
Keywords: IBS, FMRI, MBSR
MeSH Terms: conditions — Irritable Bowel Syndrome; Ichthyosis Bullosa of Siemens | interventions — Mindfulness

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- mindfulness treatment (Experimental): Mindfulness based stress reduction is the intervention in this single arm trial
  Interventions: Behavioral: Mindfulness based Stress Reduction Training (MBSR)

INTERVENTIONS:
Behavioral: Mindfulness based Stress Reduction Training (MBSR) — 8 (2 hr) classes weekly of MBSR and required homework of MBSR practice approximately 30 minutes per day.
  Other Names: Spastic colon; Irritable colon; MBSR; Mindfulness Meditation

SUMMARY:
The purpose of this study is to use functional magnetic resonance imaging (fMRI) to evaluate brain resting state networks, responses to abdominal stimuli and the effect of MBSR Training on these measures. The goal of this study is to identify biomarkers of IBS and assess the responsiveness these biomarkers after MBSR Training. A biomarker, or biological marker, is in general a substance or measure used as an indicator of a biological state. It is a characteristic that is measured and evaluated as an indicator of normal biological processes, disease processes, or responses to a therapeutic intervention, in this case MBSR.

DETAILED DESCRIPTION:
Irritable bowel syndrome (IBS) is the most common chronic visceral pain disorder ranking among the most common of all persistent pain disorders with prevalence rates of 8-12% of the population.3 Diagnostic criteria for IBS include persistent abdominal pain and/or discomfort associated with changes in bowel habit. In the majority of patients, symptoms of other co-morbid pain conditions, such as epigastric pain (functional dyspepsia), pelvic pain (IC/PBS) and musculoskeletal pain (FM) are reported. Estimates are that >50% of the U.S. workforce experiences some type of pain and 13% lose productive work time due to pain over a 2 week period, leading to over 60 billion dollars per year in lost productivity costs.4 There are no generally agreed upon biomarkers for IBS, and diagnoses are exclusively based on subjective symptom criteria. As with most of the persistent pain disorders, IBS patients and their providers have increasingly embraced a biopsychosocial model incorporating psychological and social factors along with physiologic factors, and this forms the basis for integrative treatment approaches. This multimodal approach often incorporates Mind-Body treatments, and there is a growing literature showing clinical efficacy in IBS for interventions incorporating such Mind-Body approaches as meditation, hypnosis, yoga and cognitive therapy.5 However, there is little understanding of the physiological mechanisms underlying mind-body therapies, and for this reason optimization of the treatments for specific individuals and populations is difficult.

In this project we aim to use neuroimaging based biomarkers of IBS to examine which of these physiological measures show changes specific to a mind-body treatment with previously documented efficacy, Mindfulness Based Stress Reduction Training or MBSR. MBSR was chosen as a target treatment for several reasons: Recent clinical trial data suggests there is efficacy in improving IBS symptoms with MBSR, it has demonstrated prior success with other chronic pain conditions and there is considerable literature on meditation associated brain changes.

The primary Objective is to validate optimal biomarker candidates by assessment of treatment responsiveness in IBS patients following Mindfulness Based Stress Reduction (MBSR). The secondary objectives are to determine the generality of optimal biomarkers from Aim 1 and 2 and look at factors such as sex, age, co-morbid pain or mood symptoms, and/or baseline disease severity as moderators of the performance of candidate biomarkers.

Also, exploratory analyses will be performed to assess the effect of an 8 week MBSR training on measures of disease cognition, quality of life and mood defined by pre and post test scores on the behavioral measures listed in the study methods.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must meet the Rome III criteria for IBS and lack red flag symptoms, such as weight loss, bloody stool, and fever. In the setting of clinical uncertainty on the part of the examining gastroenterologist, laboratory testing or prior medical records may be requested.
2. Upper gastrointestinal symptoms, ie. dyspepsia or heartburn, are acceptable as long as IBS is their most bothersome symptom complex.
3. Subject cannot have completed structured training in MBSR or other mindfulness or meditation.
4. Subject cannot be currently practicing MBSR.
5. A minimal severity score of 75 on the IBS-SSS at screening will be required to ensure at least mild-moderate symptoms at baseline.
6. Literate in English
7. Ambulatory without a need for assistive devices.
8. Able to participate in the sitting and mild yoga positions required for the MBSR course.
9. Right handed due to importance of laterality in brain imaging analysis
10. Not pregnant, nursing or postpartum.
11. No metals in body, including ferrous metallic implants and tattoos
12. No history of claustrophobia.
13. Able to lay still on back for extended period of time ( about 90 minutes).
14. if unable to participate in the MRI portion of the study you may be eligible to come to the MBSR classes at no cost if you agree to complete the classes, homework and on-line questionnaires.

Exclusion criteria:

1. Planned major medical intervention in the next 6 months (e.g. surgery), or surgery in the past 6 months.
2. Presence of a significant and ongoing medical problem that would interfere with participation in the study or testing the study hypotheses (e.g. major heart disease, neurological disorders, inflammatory bowel disease, etc).
3. Presence of a major psychiatric diagnosis such as schizophrenia, Bipolar disorder, Post-traumatic Stress Disorder, or Obsessive Compulsive disorder. However, subjects with a history of DSMIV diagnosis of Anxiety or Depression, in whom symptoms are not active will be allowed but noted for post-hoc analysis.
4. use of centrally acting medications that will interfere with the neuroimaging testing (e.g. narcotic medications). As in past studies we will allow subjects taking stable doses of antidepressant medications (TCAs, SSRIs, SNRIs) for at least six months prior to study to participate.
5. Body Mass Index greater than 30.
6. Current or past history of chronic pain syndrome other than IBS in the IBS group (pain >6 months at any location).
7. History of gastrointestinal surgery other than uncomplicated appendectomy or cholecystectomy.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 119 (Actual)
Dates: Start 2013-01; Primary Completion 2016-03-20 (Actual); Study Completion 2018-03-20 (Actual)

PRIMARY OUTCOMES:
Validate Optimal Biomarker candidates | After MBSR training (8 weeks).
  To validate optimal brain biomarker candidates by assessment of treatment responsiveness in IBS patients following and 8 week course in Mindfulness Based Stress Reduction (MBSR).

SECONDARY OUTCOMES:
Specificity, generality and moderation of biomarker response to MBSR treatment. | Post MBSR training at 3 month follow up.
  Specificity of biomarker response to MBSR measured by changes in selected biomarker candidates correlation w/improvement in mindfulness at end of treatment & 3-month f/u.
  Determine generality of optimal biomarkers via examination of factors such as sex, age, co-morbid pain,mood, and/or baseline disease severity, as moderators of biomarker performance.
  Moderation of biomarker performance by symptoms: Disease severity, duration, and comorbid symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Kirsten Tillisch, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- Oppenheimer Center for Neurobiology of Stress, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Neuroimaging data will be shared after initial analysis and publication at pain.ucla.edu to members of the Pain repository